CLINICAL TRIAL: NCT00645346
Title: A Phase I, Randomized, Single-blind, Controlled, Single Center Study to Evaluate the Safety and Immunogenicity of a Dose Range of Glycoconjugate Antigen Vaccine of Group B Streptococcus in Healthy Women 18- 40 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Novartis Vaccines and Diagnostics s.r.l., Novartis
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V98P2
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Invasive Group B Streptococcus (GBS) Disease
Keywords: GBS
MeSH Terms: conditions — Guillain-Barre Syndrome; Disease

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Subjects will receive either 5, 10 or 20 mcg of the vaccine
  Interventions: Biological: GBS glycoconjugate vaccine
- 2 (Placebo Comparator): Subjects will receive placebo control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBS glycoconjugate vaccine — Study subjects will receive either GBS conjugate vaccine or placebo. Total study size is 65. Study subjects will be followed for a total of 12 months after their last vaccination.
  Arms: 1
Biological: Placebo — Subjects will receive one dose of placebo
  Arms: 2

SUMMARY:
The goals of the proposed study are to evaluate the safety, tolerability and immunogenicity of a GBS vaccine. Previous studies suggest that immune responses against GBS can protect humans from infection.

ELIGIBILITY:
Inclusion Criteria:

* healthy females 18 through 40 years of age;
* have provided written informed consent after the nature of the study has been explained;
* are available for all visits scheduled for the study (i.e. are not planning to leave the area before the end of the study period);
* are in good health as determined by: medical history ,physical assessment

Exclusion Criteria:

* unwilling or unable to give written informed consent to participate in the study;
* pregnant (serum pregnancy test)
* unwilling to use acceptable birth control from screening and until at least 3 months after the final immunization
* nursing (breastfeeding) mothers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of an intramuscular GBS conjugate vaccine | 1 month

SECONDARY OUTCOMES:
To study the magnitude and durability of GBS-specific antibody responses over 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Institute for Pharmacokinetic and Analytical Studies I.P.A.S., Ligornetto, Ligornetto, Switzerland